CLINICAL TRIAL: NCT04071262
Title: A Phase 1 Study of Abemaciclib in Combination With Other Anti-Cancer Therapy in Japanese Patients With Advanced Cancer
Brief Title: A Study of Abemaciclib (LY2835219) in Combination With Other Anti-Cancer Therapies in Japanese Participants With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17229; I3Y-JE-JPCQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09-15

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — abemaciclib; Abiraterone Acetate; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Abemaciclib + Abiraterone Acetate + Prednisolone (Experimental): Abemaciclib, abiraterone acetate and prednisolone given orally.
  Interventions: Drug: Abemaciclib; Drug: Abiraterone Acetate; Drug: Prednisolone

INTERVENTIONS:
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219
Drug: Abiraterone Acetate — Administered orally
Drug: Prednisolone — Administered orally

SUMMARY:
The purpose of this study is to see if the study drug abemaciclib in combination with other anti-cancer therapies is safe in Japanese participants with advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participant with histologically confirmed adenocarcinoma of the prostate.
* Participant with metastatic disease documented by positive bone scan and/or measurable soft tissue metastatic lesions by computed tomography (CT) or magnetic resonance imagining (MRI).
* Participant who has serum testosterone level is ≤1.73 nanomoles per liter (nmol/L) (50 nanograms per deciliter).
* Participant who has progressive disease at study entry demonstrated during continuous androgen-deprivation therapy (ADT)/post orchiectomy.
* Participant with adequate organ function.
* Participant with Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.

Exclusion Criteria:

* Participant who was treated with cytochrome P450 (CYP)17 inhibitors (including abiraterone acetate, TAK-700, TOK-001, and ketoconazole).
* Participant who was treated with abemaciclib or any cyclin dependent kinase 4 and 6 (CDK4 and 6) inhibitors.
* Participant who has prior cytotoxic chemotherapy for metastatic castration-resistant prostate cancer (mCRPC), prior radiopharmaceuticals for prostate cancer (PCa), or prior sipuleucel-T.
* Participant who has gastrointestinal disorder affecting absorption or inability to swallow large pills.
* Participant who has clinically active or chronic liver disease, moderate/severe hepatic impairment, ascites, or bleeding disorders secondary to hepatic dysfunction.
* Participant who has known or suspected central nervous system metastatic disease.
* Participant who was treated with drugs known to be strong inhibitors, or strong or moderate inducers of cytochrome P450 3A4 (CYP3A4) and the treatment cannot be discontinued or switched prior to starting study treatment.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities (DLTs) | Baseline through Cycle 1 (28 Day Cycle)
  Number of Participants with DLTs

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Time Curve (AUC) of Abemaciclib in Combination with Abiraterone Acetate plus Prednisolone | Predose Cycle 1 Day 1 through Predose Cycle 3 Day 1 (28 Day Cycles)
  PK: AUC of Abemaciclib in Combination with Abiraterone Acetate plus Prednisolone
PK: Maximum Concentration (Cmax) of Abemaciclib in Combination with Abiraterone Acetate plus Prednisolone | Predose Cycle 1 Day 1 through Predose Cycle 3 Day 1 (28 Day Cycles)
  PK: Cmax of Abemaciclib in Combination with Abiraterone Acetate plus Prednisolone

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- Japan (2):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Yokohama City University Medical Center, Yokohama, Kanagawa

IPD SHARING:
Plan to Share IPD: No